CLINICAL TRIAL: NCT03455023
Title: Impact of Individualized Pharmaceutical-care on Medication Adherence and Outcome of Cancer Pain in Opioid-tolerant Inpatients
Brief Title: Individualized Pharmaceutical-care for Inpatients With Cancer Pain
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Zhejiang Cancer Hospital (Other)
Responsible Party: Principal Investigator, Ping Huang, Chief of Pharmacy, Zhejiang Cancer Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: ECCOPG-002
Record Dates: First submitted 2018-01-30; First posted 2018-03-06 (Actual); Last update posted 2019-01-15 (Actual); Status verified 2019-01

CONDITIONS: Cancer Pain
Keywords: Cancer pain; Pharmaceutical care
MeSH Terms: conditions — Cancer Pain | interventions — Pharmaceutical Services

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- pharmaceutical care intervention group (Experimental): Patients will receive individualized pharmaceutical care in addition to usual medical care.
  Interventions: Other: pharmaceutical care
- control group (No Intervention): Patients will receive usual medical care.

INTERVENTIONS:
Other: pharmaceutical care — Patients receive pharmaceutical care including individualized evaluation and intervention of adherence, efficacy and safety in cancer pain treatment.
  Arms: pharmaceutical care intervention group

SUMMARY:
The purpose of the study is to investigate the impact of pharmaceutical care on cancer pain treatment for opioid-tolerant inpatients

DETAILED DESCRIPTION:
This study is a prospective multicenter randomized controlled study to investigate the impact of pharmaceutical care on cancer pain treatment for opioid-tolerant inpatients.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 years or older;
* Histologically confirmed solid tumor;
* Diagnosed chronic cancer pain;
* Opioid-tolerant patients;
* Overall survival is expected to be over 3 months;
* Karnofsky performance score≥50;
* Willing and able to comply with the protocol

Exclusion Criteria:

* Current pregnancy or breastfeeding;
* Patients diagnosed with non-cancer pain;
* Patients treated with patient-controlled analgesia;
* Patients with pathological fracture, gastrointestinal obstruction, severe infection, non-opioid related intractable constipation;
* Patients with mental disorder;
* Creatinine clearance rate <15mL/min;
* ALT or AST ≥ 10 fold of upper limit of normal value

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2018-06-30 (Actual); Primary Completion 2019-06-30 (Estimated); Study Completion 2019-06-30 (Estimated)

PRIMARY OUTCOMES:
Change in medication adherence | Change from baseline at 1 month after discharge
  The investigators will measure the change in medication adherence via Morisky Scale. Morisky Scale contains 4 questions, and the total score ranges from 0 to 4 with lower scores indicating higher adherence.

SECONDARY OUTCOMES:
Change in pain score | Change from baseline at 1 month after discharge
  Comparison of pain score of cancer pain patients with or without pharmaceutical care. Pain score will be assessed using numeric rating scale (NRS). An NRS allows a person to describe the intensity of his/her pain as a number usually ranging from 0 to 10, where "0" means "no pain" and "10" means pain as "bad as it could be."
Change in quality of life | Change from baseline at 1 month after discharge
  Comparison of quality of life of cancer pain patients with or without pharmaceutical care. Quality of life is assessed using EuroQol- 5 Dimension (EQ-5D). It is a questionnaire to measure quality of life. It contains 5 domains: Mobility; Self-care; Usual activity; Pain; Anxiety/depression. It also contains a visual analogue scale. Weights are used to score the responses to the 5 domains, with scores ranging from 0 to 1 (where a score of 1 represents a perfect state). For the visual analogue scale, participants draw a line from a box to the point on the thermometer-like scale corresponding to their health state, 0-100 (100 = Best health state)
Change in patients' knowledge of cancer pain and analgesics | Change from baseline at 1 month after discharge
  Comparison of knowledge of cancer pain and analgesics for cancer pain patients with or without pharmaceutical care. Knowledge of pain treatment and analgesics will be assessed using investigator designed questionnaire. This questionnaire consists of 16 items assessing patients' knowledge about cancer pain, treatment of cancer pain and medications for cancer pain. The total score ranges from 0 to 16 with higher score indicating better knowledge.
Incidence of adverse events [safety and tolerability] | Up to 1 month after discharge
  Adverse events will be assessed throughout the study according the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Event (CTCAE) Version 4.0. Number of subjects who experienced an adverse event in this study is presented.

CONTACTS AND LOCATIONS:
Overall Officials: Ping Huang, Doctor, Principal Investigator — Zhejiang Cancer Hospital
Locations (1):
- Zhejiang cancer hospital, Hangzhou, Zhejiang, China

REFERENCES:
- [Derived] Zheng X, Ding H, Xu S, Xie R, Liu Y, Zhai Q, Fang L, Tong Y, Sun J, Xin W, Wu N, Chen J, Shi W, Yang L, Li H, Shao J, Wang Y, Yu H, Zhang B, Du Q, Yang Y, Zhang X, Duan C, Zhao Q, Shi J, Huang J, Fan Q, Cheng H, Chen L, Kong S, Zhang H, Gong L, Zhang Y, Song Z, Yang Y, Zhou S, Huang C, Lin J, Wang C, Huang X, Wei Q, Sun Y, Huang P. Pharmacist-Led Management Improves Treatment Adherence and Quality of Life in Opioid-Tolerant Patients With Cancer Pain: A Randomized Controlled Trial. Pain Ther. 2022 Mar;11(1):241-252. doi: 10.1007/s40122-021-00342-0. Epub 2022 Jan 29. PMID 35092599